CLINICAL TRIAL: NCT05116982
Title: Interventional Study to Evaluate the Effect of Three Silicon Based Food Supplements on the Urinary Excretion of Aluminum and Other Metals. Randomized, Parallel, Controlled and Double Blind Study (SILIAL)
Brief Title: Effect of Three Silicon Based Food Supplements on the Urinary Excretion of Aluminum and Other Metals (SILIAL)
Acronym: SILIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Silicium Laboratories S.L. (Unknown); San Antonio Technologies S.L. (Unknown); Catholic University of Murcia (UCAM) (Unknown); Zaidin Experimental Station, Spanish Council for Scientific Research (CSIC) Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAT-EURECAT-01-20
Record Dates: First submitted 2021-10-08; First posted 2021-11-11 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Aluminium Overload; Biological Availability
Keywords: Silicon; Aluminum; urinary excretion; Food supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ORGONO Living Silica Acacia Gum-MMST Powder (Experimental): ORGONO Living Silica Acacia gum-MMST Power. In capsules. One capsule a day for 7 days.
  Interventions: Dietary Supplement: ORGONO Living Silica Acacia Gum-MMST Powder
- ORGONO Living Silica Malto-OSA Powder (Experimental): ORGONO Living Silica Malto-OSA Powder. In capsules. One capsule a day for 7 days.
  Interventions: Dietary Supplement: ORGONO Living Silica Malto-OSA Powder
- ORGONO Living Silica Collagen Booster (Experimental): ORGONO Living Silica Collagen Booster. Liquid. One bottle a day for 7 days.
  Interventions: Dietary Supplement: ORGONO Living Silica Collagen Booster
- Placebo (Placebo Comparator): Placebo. In capsules and liquid. One capsule and one bottle a day for 7 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ORGONO Living Silica Acacia Gum-MMST Powder — Participants will consume one capsule per day and one bottle per day. Capsule composition: Acacia Gum 336.1 mg/capsule; Monomethylsilanetriol 34.9 mg/capsule; Hydroxypropyl methylcellulose 95 mg/capsule. Bottle composition: water 100 ml. Silicon content per dose: 10.4 mg.
  Arms: ORGONO Living Silica Acacia Gum-MMST Powder
Dietary Supplement: ORGONO Living Silica Malto-OSA Powder — Participants will consume one capsule per day and one bottle per day. Capsule composition: Maltodextrin 311.4 mg/capsule; Silicic acid 35.6 mg/capsule; Hydroxypropyl methylcellulose 95 mg/capsule. Bottle composition: water 100 ml. Silicon content per dose: 10.4 mg.
  Arms: ORGONO Living Silica Malto-OSA Powder
Dietary Supplement: ORGONO Living Silica Collagen Booster — Participants will consume one capsule per day and one bottle per day. Capsule composition: Hydroxypropyl methylcellulose 320 mg/capsule. Bottle composition: water 99.9646 g/100 ml; Silicic acid 23.65 mg/100 ml; Monomethylsilanetriol 11.75 mg/100 ml. Silicon content per dose: 10.4 mg.
  Arms: ORGONO Living Silica Collagen Booster
Dietary Supplement: Placebo — Participants will consume one capsule per day and one bottle per day. Capsule composition: Hydroxypropyl methylcellulose 320 mg/capsule. Bottle composition: water 100 ml.
  Arms: Placebo

SUMMARY:
Aluminum is a very abundant element in nature. Humans are exposed to this metal through the environment, diet, and drinking water, as well as through the consumption of certain medications.

Aluminum is not an essential element for human, being able to become neurotoxic when it reaches the brain once ingested at very high doses and, above all, if there is also kidney dysfunction.

Silicon is one of the most abundant elements on the planet and although it is not considered an essential element for humans, some beneficial activities have been documented.

Silicon has been found to be readily available in food and that 41% of ingested silicon is excreted in the urine, with a significant correlation between silicon ingested with food and urinary silicon excretion.

The most bioavailable silicon is that found in the form of silicic acid or orthosilicic acid.

Numerous studies suggest that silicon can reduce the oral absorption of aluminum and / or improve its excretion and, therefore, protect against the adverse effects induced by the ingestion of aluminum.

In a clinical study with healthy individuals as a control group for Alzheimer's disease, the levels of aluminum excretion were analyzed after the continuous ingestion of water enriched in silicon. The results in the first urine of the morning during the first week of ingestion of the enriched water showed that the excretion of aluminum was 136.9 ± 81.4 µmol / nmol creatinine while in the baseline week it was lower, 98.8 ± 64.3 nmol / nmol creatinine. These results indicated that the Al excreted came from Al stored in the body.

The main objective of the study is to evaluate the effect of the consumption of three food supplements formulated with different silicon compounds (monomethylsilanetriol and / or silicic acid) on the urinary excretion of aluminum.

The secondary objectives of the study are to evaluate:

* the bioavailability of the silicon contained in three food supplements formulated with different silicon compounds.
* the effect of the consumption of three food supplements formulated with different silicon compounds on urinary excretion of mercury, nickel, arsenic, cadmium, iron and copper.
* the safety of the consumption of three food supplements formulated with different silicon compounds.

DETAILED DESCRIPTION:
It will be conducted a single-center, randomized, controlled, double-blind clinical trial with four groups in parallel (placebo, Supplement A, Supplement B and Supplement C).

The study will be carried out with a total of 40 individuals (10 individuals per group), men and women aged 40 to 65 years. Individuals will have normal serum creatinine levels: up to 1.1mg/dl in women and up to 1.4mg/dl in men.

The investigational products involved in this study are four food supplements made from silicon compounds and the corresponding placebos.

Each participant will receive a kit containing a bottle with 10 capsules and a bottle of 100 ml of liquid according to the treatments corresponding to the randomly assigned group.

During the study, the volunteers will consume one capsule and 100ml of product each day for 7 days. The first morning urine will be collected during the 7 days of treatment and also during the previous 7 days to analyze the baseline values. In addition, on days 6 and 7 of the study, the urine will be collected in three fractions up to 24h to evaluate the bioavailability of silicon.

Participants will make a total of 5 visits, including the pre-selection visit. In these visits, the following will be carried out: Revision of Inclusion and exclusion criteria; Informed consent signature;Safety biochemistry; Demographic variables (age, sex), anthropometric variables; Evaluation of dietary intake; Randomization; Delivery of the sampling material; Verification of compliance with dietary requirements; Collection of urine samples; Investigation product delivery; Determination of metals in urine; Registration of Medication and food supplements; concomitants adverse event registry.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 to 65.
* Individuals with normal serum creatinine levels: up to 1.1 mg/dl in women and up to 1.4 mg/dl in men.

Exclusion Criteria:

* Individuals taking any type of medication and/or supplement containing aluminum, including antacids.
* Individuals who take food supplements and/or medication that contains mercury, nickel, arsenic, cadmium, iron, copper, and silicon.
* Individuals who eat mineral-enriched foods.
* Individuals allergic to any component of the dietary supplements of the study.
* Individuals with urge, stress or mixed urinary incontinence. Involuntary loss of urine accompanied by symptoms of both urge or stress urinary incontinence diagnosed by your primary care physician. In case of absence of diagnosis, the IU-4 questionnaire will be carried out.
* Pregnancy or breastfeeding.
* Individuals with any chronic gastrointestinal disease.
* Individuals with chronic kidney disease (or serum creatinine levels ≥ 1.7 mg/dl in men and ≥ 1.5 mg/dl in women).
* Be participating or have participated in a clinical trial or study of nutritional intervention in the last 30 days before study inclusion.
* Being a smoker.
* Consume 2 or more Standard Beverage Units daily or 17 weekly in women, or consume 4 or more Standard Beverage Units daily or 28 weekly in mens.
* Individuals whose condition does not allow them to carry out the study procedures strictly.
* Individuals with diseases with manifest symptoms that may influence the objectives of the study.
* Individuals with BMI≥ 30 kg/m^2.
* Individuals whose consumption of foods rich in silicon, aluminum, mercury, nickel, arsenic, cadmium, iron and copper are high.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of aluminum | 7 days
  Aluminum levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary aluminum levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of aluminium will be calculated by means of the average excreted levels of aluminium in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Aluminum levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.

SECONDARY OUTCOMES:
Bioavailability of silicon | 24 hours
  The bioavailability of silicon will be calculated by urine silicon concentration. Silicon levels will be determined in three fractions of time (8:30-11:30 hours; 11:30-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement. Silicon bioavailability will be calculated by the difference in the sum of silicon levels in all urine fractions before and after consumption of each silicon supplement. Silicon levels in urine will be measured by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by volume of urine.
Urinary excretion of mercury | 7 days
  Mercury levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary mercury levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of mercury will be calculated by means of the average excreted levels of mercury in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Mercury levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.
Urinary excretion of nickel | 7 days
  Nickel levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary nickel levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of nickel will be calculated by means of the average excreted levels of nickel in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Nickel levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.
Urinary excretion of arsenic | 7 days
  Arsenic levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary arsenic levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of arsenic will be calculated by means of the average excreted levels of arsenic in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Arsenic levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.
Urinary excretion of cadmium | 7 days
  Cadmium levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary cadmium levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of cadmium will be calculated by means of the average excreted levels of cadmium in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Cadmium levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.
Urinary excretion of iron | 7 days
  Iron levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary iron levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of iron will be calculated by means of the average excreted levels of iron in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Iron levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.
Urinary excretion of copper | 7 days
  Copper levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary copper levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively. Urinary excretion of copper will be calculated by means of the average excreted levels of copper in urine for 7 days and considering the difference between the levels excreted in urine before and after the consumption of each silicon supplement.
  Copper levels in urine will be quantified by Inductively Coupled Plasma-Optical Emission Spectrometry and will be expressed by mmol of excreted creatinine.
Urinary levels of creatinine | 14 days
  Creatinine levels in the first morning urine will be determined before consuming the dietary supplement every day for 6 days and after consuming the dietary supplement every day for 6 days. Furthermore, at days 6th and 7th urinary creatinine levels will be determined in three fractions of time (8:30-11:30 hours; 11:30h-14:30 hours; 14:30-24 hours) before and after consumption of the dietary supplement, respectively.
  Creatinine levels in urine will be quantified by a colorimetric kit.
Security | 7 days
  The safety of the dietary supplements will be evaluated through the analysis of renal markers (urea and creatinine), liver markers (transaminases) and blood count at pre-selection visit and after the consumption of the silicon supplement for 7 days. To measure the security of each silicon supplement, results obtained after each silicon supplement ingestion will be compared with results obtained before its consumption.
Adverse events | Every day for 14 days
  Adverse events will be recorded throughout the study from the initial visit to the final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Del Bas, PhD, Study Director — UTNS (Eurecat-Reus); Pilar Zafrilla, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (2):
- Spain (2):
  - Grupo de investigación de nutrición, estrés oxidativo y biodisponibilidad. Universidad Católica de Murcia (UCAM), Guadalupe, Murcia
  - Eurecat, Reus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat-Reus. — http://eurecat.org